CLINICAL TRIAL: NCT00161174
Title: Cardiovascular Morbidity in Testicular Cancer Survivors: Study of Risk Factors and Assessment of Pharmacogenomic Determinants of Toxicity. (KWF RUG 2004-3157)
Brief Title: Cardiovascular Morbidity in Testicular Cancer Survivors: Study of Risk Factors and Assessment of Pharmacogenomic Determinants of Toxicity
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: KWF RUG 2004-3157; KWF RUG 2004-3157
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Non-seminomatous Testicular Cancer
Keywords: testicular cancer; cardiovascular morbidity; cardiovascular risk factors; pharmacogenomic determinants
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For cured patients with complete data on cardiovascular risk factors and presence of subclinical cardiovascular damage only DNA will be collected.

SUMMARY:
BACKGROUND:

Evidence has emerged that patients cured with cisplatin-bleomycin chemotherapy from disseminated testicular cancer (TC) develop a large number of cardiovascular risk factors (CRF) several years later. Recently, we observed an increased incidence of cardiac events 10-20 years after chemotherapy, possibly as a result of increased occurrence of CRF. Additional cardiovascular damage was observed after treatment: disturbed diastolic function of the left ventricle, microalbuminuria and increased endothelial damage parameters. Furthermore, a metabolic syndrome (syndrome X) with insulin-resistance, dyslipidemia, hypertension and endothelial damage was found in about one third of our cured patients. The investigators hypothesize that endothelial damage and metabolic changes caused by the bleomycin and cisplatin chemotherapy are the main causes for the observed increase in cardiovascular disease in these young cancer survivors. Genetic susceptibility may be an important determinant of individual risk of toxicity in individual patients.

PURPOSE:

1. To identify risk factors for cardiovascular disease (CVD) following testicular cancer.
2. To obtain insight into the pathway(s) of CVD development, by examining whether clinical CVD following testicular cancer is associated with a preceding unfavorable cardiovascular risk factor profile and/or with treatment-related factors.
3. To investigate genetic polymorphisms in pathogenetically important pathways that are potentially involved in the development of treatment related cardiovascular morbidity following testicular cancer.

PATIENTS AND METHODS:

Patients with non-seminomatous testicular cancer who have been uniformly treated with orchidectomy and cisplatin-bleomycin combination chemotherapy at the University Hospital Groningen, The Netherlands, since 1977 but before 2000 are eligible. 380 patients with non-seminomatous testicular cancer fulfill these criteria. A close routine follow-up of these patients after treatment has been done at the University Hospital Groningen. Clinical characteristics of these patients, treatment details including outcome and long-term follow-up are being registered systematically. From all patients who agree to participate assessment of their cardiovascular risk factors and the presence of subclinical cardiovascular damage will be performed by means of several measurement techniques. Also genomic DNA will be collected for studies on polymorphisms in pathogenetically important pathways. For the total cohort of patients several different late effects phenotypes of cardiovascular damage and cardiovascular risk factor patterns will be derived from the available data. These toxicity phenotypes will be used to select cases and controls from the total cohort to test candidate genetic polymorphisms on their association with occurrence of toxicity. The association of the different genetic polymorphisms with the toxicity phenotype will be estimated by comparing cases with different toxicity phenotypes with controls without that phenotype.

POSSIBLE RESULTS This research will provide insight into the pathogenesis of cardiovascular disease after treatment for testicular cancer. The main outcome will be the possibility to select individually those patients who are likely to have an increased risk to encounter specific cardiovascular toxicity during or after chemotherapy treatment for TC. This will provide opportunities for the tailoring of potential toxic treatment and/or guide primary and secondary prevention strategies for serious side effects of chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-seminomatous testicular cancer
* Have been uniformly treated with orchidectomy and cisplatin-bleomycin combination chemotherapy at the University Hospital Groningen, The Netherlands, since 1977 but before 01-01-2000 are eligible.

Exclusion Criteria:

* N/A

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with non-seminomatous testicular cancer who have been uniformly treated with orchidectomy and cisplatin-bleomycin combination chemotherapy
Sampling Method: Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2005-07; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth G.E. de Vries, MD, PhD, Study Director — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands

REFERENCES:
- [Background] Einhorn LH. Treatment of testicular cancer: a new and improved model. J Clin Oncol. 1990 Nov;8(11):1777-81. doi: 10.1200/JCO.1990.8.11.1777. PMID 1700077
- [Background] Stoter G, Koopman A, Vendrik CP, Struyvenberg A, Sleyfer DT, Willemse PH, Schraffordt Koops H, van Oosterom AT, ten Bokkel Huinink WW, Pinedo HM. Ten-year survival and late sequelae in testicular cancer patients treated with cisplatin, vinblastine, and bleomycin. J Clin Oncol. 1989 Aug;7(8):1099-104. doi: 10.1200/JCO.1989.7.8.1099. PMID 2474060
- [Background] Meijer S, Sleijfer DT, Mulder NH, Sluiter WJ, Marrink J, Koops HS, Brouwers TM, Oldhoff J, van der Hem GK, Mandema E. Some effects of combination chemotherapy with cis-platinum on renal function in patients with nonseminomatous testicular carcinoma. Cancer. 1983 Jun 1;51(11):2035-40. doi: 10.1002/1097-0142(19830601)51:113.0.co;2-8. PMID 6340821
- [Background] Hansen SW, Groth S, Daugaard G, Rossing N, Rorth M. Long-term effects on renal function and blood pressure of treatment with cisplatin, vinblastine, and bleomycin in patients with germ cell cancer. J Clin Oncol. 1988 Nov;6(11):1728-31. doi: 10.1200/JCO.1988.6.11.1728. PMID 2460594
- [Background] Roth BJ, Greist A, Kubilis PS, Williams SD, Einhorn LH. Cisplatin-based combination chemotherapy for disseminated germ cell tumors: long-term follow-up. J Clin Oncol. 1988 Aug;6(8):1239-47. doi: 10.1200/JCO.1988.6.8.1239. PMID 2457658
- [Background] Vogelzang NJ, Torkelson JL, Kennedy BJ. Hypomagnesemia, renal dysfunction, and Raynaud's phenomenon in patients treated with cisplatin, vinblastine, and bleomycin. Cancer. 1985 Dec 15;56(12):2765-70. doi: 10.1002/1097-0142(19851215)56:123.0.co;2-2. PMID 2413982
- [Background] Boyer M, Raghavan D, Harris PJ, Lietch J, Bleasel A, Walsh JC, Anderson S, Tsang CS. Lack of late toxicity in patients treated with cisplatin-containing combination chemotherapy for metastatic testicular cancer. J Clin Oncol. 1990 Jan;8(1):21-6. doi: 10.1200/JCO.1990.8.1.21. PMID 1688614
- [Background] Doll DC, List AF, Greco FA, Hainsworth JD, Hande KR, Johnson DH. Acute vascular ischemic events after cisplatin-based combination chemotherapy for germ-cell tumors of the testis. Ann Intern Med. 1986 Jul;105(1):48-51. doi: 10.7326/0003-4819-105-1-48. PMID 2424354
- [Background] Samuels BL, Vogelzang NJ, Kennedy BJ. Severe vascular toxicity associated with vinblastine, bleomycin, and cisplatin chemotherapy. Cancer Chemother Pharmacol. 1987;19(3):253-6. doi: 10.1007/BF00252982. PMID 2438065
- [Background] Vogelzang NJ, Frenning DH, Kennedy BJ. Coronary artery disease after treatment with bleomycin and vinblastine. Cancer Treat Rep. 1980 Oct-Nov;64(10-11):1159-60. No abstract available. PMID 6161700
- [Background] Gerl A, Clemm C, Wilmanns W. Acute cerebrovascular event after cisplatin-based chemotherapy for testicular cancer. Lancet. 1991 Aug 10;338(8763):385-6. doi: 10.1016/0140-6736(91)90521-p. No abstract available. PMID 1677724
- [Background] Nichols CR, Roth BJ, Williams SD, Gill I, Muggia FM, Stablein DM, Weiss RB, Einhorn LH. No evidence of acute cardiovascular complications of chemotherapy for testicular cancer: an analysis of the Testicular Cancer Intergroup Study. J Clin Oncol. 1992 May;10(5):760-5. doi: 10.1200/JCO.1992.10.5.760. PMID 1285740
- [Background] Gietema JA, Sleijfer DT, Willemse PH, Schraffordt Koops H, van Ittersum E, Verschuren WM, Kromhout D, Sluiter WJ, Mulder NH, de Vries EG. Long-term follow-up of cardiovascular risk factors in patients given chemotherapy for disseminated nonseminomatous testicular cancer. Ann Intern Med. 1992 May 1;116(9):709-15. doi: 10.7326/0003-4819-116-9-709. PMID 1558341
- [Background] Gietema JA, de Vries EG, Sleijfer DT. Increased incidence of cardiovascular risk factors in cured testicular cancer patients. J Clin Oncol. 1992 Oct;10(10):1652. No abstract available. PMID 1328550
- [Background] Boyer M, Raghavan D. Toxicity of treatment of germ cell tumors. Semin Oncol. 1992 Apr;19(2):128-42. PMID 1313191
- [Background] Raghavan D, Cox K, Childs A, Grygiel J, Sullivan D. Hypercholesterolemia after chemotherapy for testis cancer. J Clin Oncol. 1992 Sep;10(9):1386-9. doi: 10.1200/JCO.1992.10.9.1386. PMID 1325540
- [Background] Bokemeyer C, Berger CC, Kuczyk MA, Schmoll HJ. Evaluation of long-term toxicity after chemotherapy for testicular cancer. J Clin Oncol. 1996 Nov;14(11):2923-32. doi: 10.1200/JCO.1996.14.11.2923. PMID 8918489
- [Background] Berger CC, Bokemeyer C, Schneider M, Kuczyk MA, Schmoll HJ. Secondary Raynaud's phenomenon and other late vascular complications following chemotherapy for testicular cancer. Eur J Cancer. 1995 Dec;31A(13-14):2229-38. doi: 10.1016/0959-8049(95)00460-2. PMID 8652248
- [Background] Hansen SW, Olsen N. Raynaud's phenomenon in patients treated with cisplatin, vinblastine, and bleomycin for germ cell cancer: measurement of vasoconstrictor response to cold. J Clin Oncol. 1989 Jul;7(7):940-2. doi: 10.1200/JCO.1989.7.7.940. PMID 2472472
- [Background] Meinardi MT, Gietema JA, van der Graaf WT, van Veldhuisen DJ, Runne MA, Sluiter WJ, de Vries EG, Willemse PB, Mulder NH, van den Berg MP, Koops HS, Sleijfer DT. Cardiovascular morbidity in long-term survivors of metastatic testicular cancer. J Clin Oncol. 2000 Apr;18(8):1725-32. doi: 10.1200/JCO.2000.18.8.1725. PMID 10764433
- [Background] Meinardi MT, Gietema JA, Van der Graaf WTA et al. Long-term vascular and metabolic sequelae of chemotherapy for metastatic testicular cancer. A comparison with long-term survivors of stage I disease. PROC ASCO 2000; 19: 331a.
- [Background] Huddart RA, Norman A, Shahidi M, Horwich A, Coward D, Nicholls J, Dearnaley DP. Cardiovascular disease as a long-term complication of treatment for testicular cancer. J Clin Oncol. 2003 Apr 15;21(8):1513-23. doi: 10.1200/JCO.2003.04.173. PMID 12697875
- [Background] Travis LB, Curtis RE, Storm H, Hall P, Holowaty E, Van Leeuwen FE, Kohler BA, Pukkala E, Lynch CF, Andersson M, Bergfeldt K, Clarke EA, Wiklund T, Stoter G, Gospodarowicz M, Sturgeon J, Fraumeni JF Jr, Boice JD Jr. Risk of second malignant neoplasms among long-term survivors of testicular cancer. J Natl Cancer Inst. 1997 Oct 1;89(19):1429-39. doi: 10.1093/jnci/89.19.1429. PMID 9326912
- [Background] Vogelzang NJ, Bosl GJ, Johnson K, Kennedy BJ. Raynaud's phenomenon: a common toxicity after combination chemotherapy for testicular cancer. Ann Intern Med. 1981 Sep;95(3):288-92. doi: 10.7326/0003-4819-95-3-288. PMID 6168223
- [Background] Yudkin JS, Forrest RD, Jackson CA. Microalbuminuria as predictor of vascular disease in non-diabetic subjects. Islington Diabetes Survey. Lancet. 1988 Sep 3;2(8610):530-3. doi: 10.1016/s0140-6736(88)92657-8. PMID 2900920
- [Background] Ross R. The pathogenesis of atherosclerosis: a perspective for the 1990s. Nature. 1993 Apr 29;362(6423):801-9. doi: 10.1038/362801a0. PMID 8479518
- [Background] Pedrinelli R, Giampietro O, Carmassi F, Melillo E, Dell'Omo G, Catapano G, Matteucci E, Talarico L, Morale M, De Negri F, et al. Microalbuminuria and endothelial dysfunction in essential hypertension. Lancet. 1994 Jul 2;344(8914):14-8. doi: 10.1016/s0140-6736(94)91047-2. PMID 7912295
- [Background] Reaven GM. Banting lecture 1988. Role of insulin resistance in human disease. Diabetes. 1988 Dec;37(12):1595-607. doi: 10.2337/diab.37.12.1595. PMID 3056758
- [Background] Talvensaari KK, Lanning M, Tapanainen P, Knip M. Long-term survivors of childhood cancer have an increased risk of manifesting the metabolic syndrome. J Clin Endocrinol Metab. 1996 Aug;81(8):3051-5. doi: 10.1210/jcem.81.8.8768873.
- [Background] Taskinen M, Saarinen-Pihkala UM, Hovi L, Lipsanen-Nyman M. Impaired glucose tolerance and dyslipidaemia as late effects after bone-marrow transplantation in childhood. Lancet. 2000 Sep 16;356(9234):993-7. doi: 10.1016/S0140-6736(00)02717-3. PMID 11041401
- [Background] Nord C, Fossa SD, Egeland T. Excessive annual BMI increase after chemotherapy among young survivors of testicular cancer. Br J Cancer. 2003 Jan 13;88(1):36-41. doi: 10.1038/sj.bjc.6600714. PMID 12556956
- [Background] Gietema JA, Meinardi MT, van der Graaf WT, Sleijfer DT. Syndrome X in testicular-cancer survivors. Lancet. 2001 Jan 20;357(9251):228-9. doi: 10.1016/S0140-6736(05)71326-X. No abstract available. PMID 11213121
- [Background] Gietema JA, Meinardi MT, Messerschmidt J, Gelevert T, Alt F, Uges DR, Sleijfer DT. Circulating plasma platinum more than 10 years after cisplatin treatment for testicular cancer. Lancet. 2000 Mar 25;355(9209):1075-6. doi: 10.1016/s0140-6736(00)02044-4. PMID 10744098
- [Background] Evans WE, Relling MV. Pharmacogenomics: translating functional genomics into rational therapeutics. Science. 1999 Oct 15;286(5439):487-91. doi: 10.1126/science.286.5439.487. PMID 10521338
- [Background] Evans WE, McLeod HL. Pharmacogenomics--drug disposition, drug targets, and side effects. N Engl J Med. 2003 Feb 6;348(6):538-49. doi: 10.1056/NEJMra020526. No abstract available. PMID 12571262
- [Background] Weinshilboum R. Inheritance and drug response. N Engl J Med. 2003 Feb 6;348(6):529-37. doi: 10.1056/NEJMra020021. No abstract available. PMID 12571261
- [Background] Vaughn DJ, Meadows AT. Cancer survivorship research: the best is yet to come. J Clin Oncol. 2002 Feb 15;20(4):888-90. doi: 10.1200/JCO.2002.20.4.888. No abstract available. PMID 11844806
- [Background] Celermajer DS, Sorensen KE, Gooch VM, Spiegelhalter DJ, Miller OI, Sullivan ID, Lloyd JK, Deanfield JE. Non-invasive detection of endothelial dysfunction in children and adults at risk of atherosclerosis. Lancet. 1992 Nov 7;340(8828):1111-5. doi: 10.1016/0140-6736(92)93147-f. PMID 1359209
- [Background] Celermajer DS, Sorensen KE, Georgakopoulos D, Bull C, Thomas O, Robinson J, Deanfield JE. Cigarette smoking is associated with dose-related and potentially reversible impairment of endothelium-dependent dilation in healthy young adults. Circulation. 1993 Nov;88(5 Pt 1):2149-55. doi: 10.1161/01.cir.88.5.2149. PMID 8222109
- [Background] La Rovere MT, Bigger JT Jr, Marcus FI, Mortara A, Schwartz PJ. Baroreflex sensitivity and heart-rate variability in prediction of total cardiac mortality after myocardial infarction. ATRAMI (Autonomic Tone and Reflexes After Myocardial Infarction) Investigators. Lancet. 1998 Feb 14;351(9101):478-84. doi: 10.1016/s0140-6736(97)11144-8. PMID 9482439
- [Background] Lefrandt JD, Hoogenberg K, van Roon AM, Dullaart RP, Gans RO, Smit AJ. Baroreflex sensitivity is depressed in microalbuminuric Type I diabetic patients at rest and during sympathetic manoeuvres. Diabetologia. 1999 Nov;42(11):1345-9. doi: 10.1007/s001250051448. PMID 10550419
- [Background] Innocenti F, Ratain MJ. Update on pharmacogenetics in cancer chemotherapy. Eur J Cancer. 2002 Mar;38(5):639-44. doi: 10.1016/s0959-8049(01)00434-8. PMID 11916544
- [Background] Sekine I, Saijo N. Polymorphisms of metabolizing enzymes and transporter proteins involved in the clearance of anticancer agents. Ann Oncol. 2001 Nov;12(11):1515-25. doi: 10.1023/a:1013164013375. PMID 11822749
- [Background] Tuimala J, Szekely G, Gundy S, Hirvonen A, Norppa H. Genetic polymorphisms of DNA repair and xenobiotic-metabolizing enzymes: role in mutagen sensitivity. Carcinogenesis. 2002 Jun;23(6):1003-8. doi: 10.1093/carcin/23.6.1003. PMID 12082022
- [Background] Libura J, Bettens F, Radkowski A, Tiercy JM, Piguet PF. Risk of chemotherapy-induced pulmonary fibrosis is associated with polymorphic tumour necrosis factor-a2 gene. Eur Respir J. 2002 May;19(5):912-8. doi: 10.1183/09031936.02.00238102. PMID 12030733
- [Background] Montoya SE, Ferrell RE, Lazo JS. Genomic structure and genetic mapping of the human neutral cysteine protease bleomycin hydrolase. Cancer Res. 1997 Oct 1;57(19):4191-5. PMID 9331073
- [Background] Montoya SE, Aston CE, DeKosky ST, Kamboh MI, Lazo JS, Ferrell RE. Bleomycin hydrolase is associated with risk of sporadic Alzheimer's disease. Nat Genet. 1998 Mar;18(3):211-2. doi: 10.1038/ng0398-211. No abstract available. PMID 9500538
- [Background] Boekholdt SM, Bijsterveld NR, Moons AH, Levi M, Buller HR, Peters RJ. Genetic variation in coagulation and fibrinolytic proteins and their relation with acute myocardial infarction: a systematic review. Circulation. 2001 Dec 18;104(25):3063-8. doi: 10.1161/hc5001.100793. PMID 11748101
- [Background] Yamada Y, Izawa H, Ichihara S, Takatsu F, Ishihara H, Hirayama H, Sone T, Tanaka M, Yokota M. Prediction of the risk of myocardial infarction from polymorphisms in candidate genes. N Engl J Med. 2002 Dec 12;347(24):1916-23. doi: 10.1056/NEJMoa021445. PMID 12477941
- [Background] Nicaud V, Raoux S, Poirier O, Cambien F, O'Reilly DS, Tiret L. The TNF alpha/G-308A polymorphism influences insulin sensitivity in offspring of patients with coronary heart disease: the European Atherosclerosis Research Study II. Atherosclerosis. 2002 Apr;161(2):317-25. doi: 10.1016/s0021-9150(01)00648-7. PMID 11888514
- [Background] Makridakis NM, di Salle E, Reichardt JK. Biochemical and pharmacogenetic dissection of human steroid 5 alpha-reductase type II. Pharmacogenetics. 2000 Jul;10(5):407-13. doi: 10.1097/00008571-200007000-00004. PMID 10898110
- [Background] Garte S. Metabolic susceptibility genes as cancer risk factors: time for a reassessment? Cancer Epidemiol Biomarkers Prev. 2001 Dec;10(12):1233-7. PMID 11751439
- [Background] Lenz HJ. The use and development of germline polymorphisms in clinical oncology. J Clin Oncol. 2004 Jul 1;22(13):2519-21. doi: 10.1200/JCO.2004.04.900. Epub 2004 Jun 1. No abstract available. PMID 15173210